CLINICAL TRIAL: NCT02829294
Title: Evaluation of a Novel Product for the Removal of Impacted Human Cerumen (Earwax)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Joseph Griffin (Industry)
Responsible Party: Sponsor-Investigator, Dr. Joseph Griffin, Chief Scientific Officer, Eosera Inc
Organization: Eosera Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOS-002
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cerumen Impaction of Both Ears

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): E002 - cerumen removal aid will be placed into the ear canal of enrolled subjects for 15 to 30 minutes
  Interventions: Device: E002 - cerumen removal aid

INTERVENTIONS:
Device: E002 - cerumen removal aid — topical treatment

SUMMARY:
This is a prospective, open-labeled clinical trial. Subjects that qualify for enrollment and provide informed consent will be treated with a novel topical cerumen (earwax) removal product. The primary goal of this pilot study is to gain an understanding of the safety and efficacy of this novel product.

DETAILED DESCRIPTION:
This is a single center, single-arm, open-label trial. Approximately 30 evaluable ears will be enrolled that have at least 50% cerumen impaction. All ears/subjects will receive at least a single dose (approximately 1 - 2 mL) of the test product applied topically in the study ear canal. The test product will be supplied from a qualified compounding pharmacy that receives a by-subject prescription from the investigator. The subject will be dosed with the head tilted in order to keep the test product in the ear canal for 15 minutes. At 5 and 10 minutes, subjects will be instructed to move their jaw up and down (and side to side) a few times and, manipulate/massage the ear canal by pressing between jawbone and ear lobe with a rotating motion for 10 seconds, which may aid in distribution of the test product in the ear canal. Fifteen minutes after product instillation, it will be removed by having the subject tilt the head over a disposable container to catch the solution. The ear canal will be irrigated (low pressure) with warm water and, the evaluator will try to visualize the tympanic membrane using an otoscope (before and after lavage). The amount (change in area, volume and depth) of the tympanic membrane that can be visualized and the categorization of cerumen impaction (according to a 5 point scale) is the primary efficacy parameter of this study. Efficacy will also be assessed using subjective questions (improvement and change in symptoms) that will be asked by the study staff and documented prior to the subject having any knowledge of the otoscope results (visualization of TP).

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females ≥ 40 years of age at enrollment;
2. Presence of excessive or impacted cerumen [excessive or impacted cerumen is identified as causing partial (> 50%) or complete occlusion of at least one ear canal when attempting to visualize the tympanic membrane];
3. Willingness to participate in the study; or
4. Mental aptitude to provide verbal and/or written informed consent without the aid of another.

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study (has been accustomed to birth control and will continue it up to and including Visit 2);
2. Presence of a tympanostomy tube at any time during the previous 12 months;
3. Presence of a non-intact tympanic membrane (TM);
4. Presence of a known or suspected ear infection;
5. Presence of known or suspected mastoiditis;
6. Use of any ototopical drug or OTC product or earwax-removal product (with the exception of water or physiologic saline) during the preceding 3 days; or
7. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data (e.g. ear eczema or seborrhea).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Griffin, PhD, Study Director — Eosera Inc
Locations (1):
- Legacy Medical Village, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fullington D, Song J, Gilles A, Guo X, Hua W, Anderson CE, Griffin J. Evaluation of the safety and efficacy of a novel product for the removal of impacted human cerumen. BMC Ear Nose Throat Disord. 2017 Jun 2;17:5. doi: 10.1186/s12901-017-0038-8. eCollection 2017. PMID 28588421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were recruited from the normal clinic population and based on the investigators prior knowledge of treating subjects with the conditions.
Pre-assignment Details: Subjects were pre-screened. If subjects agreed to participate, treatment was scheduled. On the treatment day, subjects were re-screened to ensure inclusion/exclusion criteria were met. Subjects were consented and then proceeded to treatment.
Groups:
- Treatment: Subjects that meet the inclusion/exclusion criteria were treated with test product per protocol
Period: Overall Study
Arm/Group | Treatment
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 19 participants and of these 19 participants there were 30 ears that individually met the inclusion criteria.
Units Other Than Participants: ears
Groups:
- Treatment: Subjects that qualify were treated per protocol
Arm/Group | Treatment
Number analyzed (Participants) | 19
Number analyzed (ears) | 30
Age, Categorical [Count of Participants; unit: Participants] — Patients greater than or equal to 40 years of age
  Participants
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Subjects were asked if they were male or female
  Participants
    Female | 4
    Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Subjects were asked to describe their ethnicity.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 18
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Symptoms related to ear wax impaction - decreased hearing, sensation of fullness, etc [Count of Participants; unit: Participants] | 7
Number of Participants with quality of life measures affected by ear wax impaction [Count of Participants; unit: Participants] — Criteria used to assess this baseline measure on Quality of Life included measures of decreased hearing, feeling of fullness in the ear, ringing or noises in the ear (tinnitus), ear itching, water trapping or cracking noise after swimming or shower, ear irritation/discomfort, earache, tingling in the ear or ear pain.
  Participants | 7
Otoscopic measurements of level of ear wax impaction [Number; unit: ears] — The level of ear wax impaction was graded using a clinical score based on how visible the tympanic membrane (ear drum) was when viewed with an otoscope as follows: A score of 1 (normal) means less than 3% of the ear drum was obstructed from view. A score of 2 (minimal) means that from 3 to 25% of the ear drum was obstructed from view by debris/ear wax. A score of 3 (mild) means that 26 to 50% of the ear drum was obstructed from view. A score of 4 (moderate) means 51 to 75% of the ear drum was obstructed from view. A score of 5 (severe) means 76-100% of the ear drum was obstructed from view. Population: The baseline measurements were taking from 19 patients. From these 19 patients, there were a total of 30 ears that met the inclusion criteria for enrollment.
  ears
    Number of ears with moderate impaction (51-75%) | 10
    Number of ears with severe impaction (76-100%) | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Ears That Showed Change in Visualization of the Tympanic Membrane (Ear Drum) Following 15 or 30 Minutes of Using the Test Product
Description: Cerumen impaction will be graded following 15 and 30 minutes after using the test product in the external ear canal. Cerumen impaction is graded by the % of the ear drum is visible using an otoscope. Grade 5 (severe) = 76-100% of the ear drum is obstructed from view. Grade 4 (moderate) = 51-75% of the ear drum is obstructed from view. Grade 3 (mild) = 26-50% of the ear drum is obstructed from view. Grade 2 = 3-25% of the ear drum is obstructed from view. Grade 1 (normal) = less than 3% of the ear drum is obstructed from view.
Time Frame: 15 and 30 minutes
Population: Individual ears that met all inclusion/exclusion criteria
Measure: Number; unit: percentage of ears
Units Other Than Participants: ears
Groups:
- Ears Treated With E002 for 1 or 2 Treatments of 15 Minutes: E002 - cerumen removal aid will be placed into the ear canal of enrolled subjects for 1 or 2 treatments of 15 minutes
  E002 - cerumen removal aid: topical treatment
Arm/Group | Ears Treated With E002 for 1 or 2 Treatments of 15 Minutes
Number analyzed (Participants) | 19
Number analyzed (ears) | 30
percentage of ears
  % of Grade 1 (normal) after 1 treatment (15 mins) | 53.3
  % of Grade 1 (normal) after 2 treatments (30 mins): number analyzed (ears) | 28
  % of Grade 1 (normal) after 2 treatments (30 mins) | 85.7

2. Primary Outcome: Safety Measured by the Collection of Unsolicited Adverse Events Reported by Patients
Description: Ear canal specific safety evaluation, measured by physician, during the course of treatment up to 48 hours post treatment and collection of adverse events (related and non-related)
Time Frame: After treatment
Population: 64.8 years +/- 12.3
Measure: Number; unit: number of ears with reported pruritus
Units Other Than Participants: ears
Groups:
- Ears Treated With E002 for 1 or 2 Treatments of 15 Minutes: Subjects that meet the inclusion/exclusion criteria were treated with test product per protocol
Arm/Group | Ears Treated With E002 for 1 or 2 Treatments of 15 Minutes
Number analyzed (Participants) | 19
Number analyzed (ears) | 30
number of ears with reported pruritus | 1

3. Secondary Outcome: Improvements in Ear Specific Clinical Symptoms After 1 or 2, 15 Minute Applications of E002
Description: Collect symptom information prior to and post treatment with the novel test solution designed to help clean and clear the ear canal of debris including cerumen
Time Frame: Immediately following 1 or 2 treatments
Population: There were 19 participants and of these 19 participants there were 30 ears that met the inclusion criteria.
Measure: Number; unit: % of participants reporting change
Groups:
- Ears Treated With E002 for 1 or 2 Treatments of 15 Minutes: Subjects with either one or 2 ears that met the inclusion/exclusion criteria were treated with test product per protocol
Arm/Group | Ears Treated With E002 for 1 or 2 Treatments of 15 Minutes
Number analyzed (Participants) | 19
% of participants reporting change
  Change in decreased hearing | 70
  Change in ear itching | 90
  Change in feelings of fullness | 90
  Change in water trapping or cracking | 80

ADVERSE EVENTS:
Time Frame: 48 hours post treatment
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=19)
Pruritis of ear (Ear and labyrinth disorders) | 1 (1) — Itching reported following treatment.

LIMITATIONS AND CAVEATS:
Single arm, open label evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less